CLINICAL TRIAL: NCT02078154
Title: Measurement of D-Dimer Levels in Patients With Confirmed Deep Vein Thrombosis
Status: Terminated | Type: Observational
Why Stopped: Decision to start a new study on DVT with another protocol
Sponsor: Diagnostica Stago (Industry)
Responsible Party: Sponsor
Other Study IDs: D-Dimer DVT
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Deep Venous Thrombosis
Keywords: D-Dimer; DVT; Wells score
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Deep Venous Thrombosis (DVT): DVT diagnosed by imaging technique with a low or moderate Wells score

SUMMARY:
Measurement of D-Di (D-Dimer) levels using the in-vitro diagnostic reagent STA® - Liatest® D-Di and STA® - Liatest® D-Di PLUS in plasma samples from patients diagnosed with Deep Vein Thrombosis (DVT) Data from this study may be used in conjunction with data from the prospective study entitled "STA® - Liatest® D-Di - Exclusion of Venous Thromboembolism (VTE)", NCT01221805, the DiET study,

ELIGIBILITY:
Inclusion Criteria:

* The study population tested will be recruited from ambulatory outpatients (presenting at the emergency unit or outpatient clinic) suspected of having DVT.
* Patient is < 80 years old.
* Patient presenting at least one of these symptoms indicative of proximal DVT: leg pain, tenderness (discomfort through palpation), leg swelling and /or edema,
* Patient has confirmed proximal DVT by imaging
* Low or moderate Wells score
* Patient provides written informed consent to participate in the sample collection

Exclusion Criteria:

* Patient presenting with a condition that may be associated with increased D-dimer levels, even in the absence of VTE, such as:

  1. Fibrinolytic therapy within the previous seven (7) days,
  2. Bone fracture or surgery (with general anesthesia longer than thirty (30) minutes) within the previous one (1) month,
  3. Deep hematoma diagnosed by imaging techniques within the previous one (1) month,
  4. Disseminated malignancies and active cancer (active cancer defined as: cancer for which therapeutic or palliative treatment is either ongoing at the time of enrolment or has stopped less than six (6) months before enrolment),
  5. Sepsis, severe infections, pneumonia within the previous 1 month,
  6. Known liver cirrhosis,
  7. Pregnancy or post-partum within the previous 1 month,
  8. Atherosclerotic vascular disease thrombosis within the previous 1month (e.g. myocardial infarction, stroke, coronary syndrome, peripheral artery disease stage III or IV),
  9. Sickle cell disease,
* Patients presenting with a suspect thrombotic event related to catheter implantation
* Ongoing therapeutic anticoagulants (curative and preventive treatment) starting twenty four (24) hours or more before the blood drawing for D-dimer testing

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proximal DVT diagnosed by imaging technique and with a low and moderate Wells score
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
STA Liatest DDi results in DVT positive cases | At the initial visit (up to 24 hours)
  Prospective, ambulatory outpatients (presenting to the emergency unit or outpatient clinic) suspected of having DVT, with a proximal positive imaging results, will be screened for eligibility using the inclusion and exclusion criteria (see Section above). Then the eligible patients will be evaluated using the Wells score and only patient with Low or moderate Pre-Test Probability (PTP) will receive full explanation concerning nature, objectives and risks associated to the participation in this study. Written informed consent will be obtained from each participating subject prior blood drawing, processing, plasma aliquoting and freezing at -80°C for D-Dimer testing (STA Liatest DDi). The whole process, starting from the moment the patient is diagnosed with DVT, should not exceed 24 hours.

SECONDARY OUTCOMES:
STA Liatest DDi Versus STA Liatest DDi Plus | At the initial visit (up to 24 hours)
  Prospective, ambulatory outpatients (presenting to the emergency unit or outpatient clinic) suspected of having DVT, with a proximal positive imaging results, will be screened for eligibility using the inclusion and exclusion criteria (see Section above). Then the eligible patients will be evaluated using the Wells score and only patient with Low or moderate PTP will receive full explanation concerning nature, objectives and risks associated to the participation in this study. Written informed consent will be obtained from each participating subject prior blood drawing, processing, plasma aliquoting and freezing at -80°C for D-Dimer testing (STA Liatest DDi Plus). The whole process, starting from the moment the patient is diagnosed with DVT, should not exceed 24 hours

OTHER OUTCOMES:
Plasma bank for DDi measurements | At the initial visit (up to 24 hours)
  Prospective, ambulatory outpatients (presenting to the emergency unit or outpatient clinic) suspected of having DVT, with a proximal positive imaging results, will be screened for eligibility using the inclusion and exclusion criteria (see Section above). Then the eligible patients will be evaluated using the Wells score and only patient with Low or moderate PTP will receive full explanation concerning nature, objectives and risks associated to the participation in this study. Written informed consent will be obtained from each participating subject prior blood drawing, processing, plasma aliquoting and freezing at -80°C for D-Dimer testing (STA Liatest DDi or STA Liatest DDi Plus to investigate unmatched results). The whole process, starting from the moment the patient is diagnosed with DVT, should not exceed 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wasan Rathbun, MD, Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States